CLINICAL TRIAL: NCT00690339
Title: Safety and Effectiveness of Style 410 Silicone-Filled Breast Implant Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan Medical (Industry)
Responsible Party: Sponsor
Organization: Allergan (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 00201; NCT00557674 (obsolete NCT alias)
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Results first posted 2014-02-04 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2013-12

CONDITIONS: Breast Augmentation; Breast Reconstruction; Revision of Augmentation or Reconstruction

ARMS (4):
- 1 (Experimental): Augmentation
  Interventions: Device: Style 410 Silicone-Filled Breast Implants
- 2 (Experimental): Reconstruction
  Interventions: Device: Style 410 Silicone-Filled Breast Implants
- 3 (Experimental): Revision-augmentation
  Interventions: Device: Style 410 Silicone-Filled Breast Implants
- 4 (Experimental): Revision-reconstruction
  Interventions: Device: Style 410 Silicone-Filled Breast Implants

INTERVENTIONS:
Device: Style 410 Silicone-Filled Breast Implants — Breast Implant Surgery

SUMMARY:
Safety and effectiveness of Style 410 Silicone-Filled Breast Implants in women undergoing primary augmentation, primary reconstruction, or revision of existing breast implants.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 18 years or older
* Patients seeking primary breast augmentation (i.e., no previous breast implant surgery) indicated for the following: Patient dissatisfaction with size or shape of breast (e.g., mammary hypoplasia), asymmetry, ptosis, aplasia
* Patients seeking breast reconstruction
* Patients seeking breast revision-augmentation
* Patients seeking breast revision-reconstruction
* Adequate tissue available to cover implants
* Patients must be willing to undergo MRI at their 1, 3, 5, 7, and 10-year follow-up visits (serial MRI). The patient must be eligible for MRI (for example, no implanted metal or metal devices and no history of severe claustrophobia that may make her ineligible for MRI).

Exclusion Criteria:

* Advanced fibrocystic disease considered to be premalignant without accompanying subcutaneous mastectomy
* Existing carcinoma of the breast, without mastectomy
* Abscess or infection in the body at the time of enrollment
* Pregnant or nursing
* Have any disease, including uncontrolled diabetes (e.g., Hb AIc > 8%), that is clinically known to impact wound healing ability
* Show tissue characteristics that are clinically incompatible with mammaplasty, such as tissue damage resulting from radiation, inadequate tissue, compromised vascularity or ulceration
* Have, or under treatment for, any condition that may constitute an unwarranted surgical risk (e.g., unstable cardiac or pulmonary problems)
* Show psychological characteristics that may be incompatible with the surgical procedure and the prosthesis, such as inappropriate attitude or motivation (e.g., body dysmorphic disorder)
* Are not willing to undergo further surgery for revision, if medically required

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 941 (Actual)
Dates: Start 2001-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Indianapolis, Indiana, United States

REFERENCES:
- [Result] Bengtson BP, Van Natta BW, Murphy DK, Slicton A, Maxwell GP; Style 410 U.S. Core Clinical Study Group. Style 410 highly cohesive silicone breast implant core study results at 3 years. Plast Reconstr Surg. 2007 Dec;120(7 Suppl 1):40S-48S. doi: 10.1097/01.prs.0000286666.29101.11. PMID 18090813
- [Result] Gladfelter J, Murphy D. Breast augmentation motivations and satisfaction: a prospective study of more than 3,000 silicone implantations. Plast Surg Nurs. 2008 Oct-Dec;28(4):170-4; quiz 175-6. doi: 10.1097/PSN.0b013e31818ea7e0. PMID 19092580
- [Result] Maxwell GP, Van Natta BW, Murphy DK, Slicton A, Bengtson BP. Natrelle style 410 form-stable silicone breast implants: core study results at 6 years. Aesthet Surg J. 2012 Aug;32(6):709-17. doi: 10.1177/1090820X12452423. Epub 2012 Jun 29. PMID 22751081
- [Result] Largent JA, Reisman NR, Kaplan HM, Oefelein MG, Jewell ML. Clinical trial outcomes of high- and extra high-profile breast implants. Aesthet Surg J. 2013 May;33(4):529-39. doi: 10.1177/1090820X13484035. Epub 2013 Apr 4. PMID 23559355
- [Result] Namnoum JD, Largent J, Kaplan HM, Oefelein MG, Brown MH. Primary breast augmentation clinical trial outcomes stratified by surgical incision, anatomical placement and implant device type. J Plast Reconstr Aesthet Surg. 2013 Sep;66(9):1165-72. doi: 10.1016/j.bjps.2013.04.046. Epub 2013 May 9. PMID 23664574

RESULTS

PARTICIPANT FLOW:
Groups:
- Augmentation: Augmentation
  Style 410 Silicone-Filled Breast Implants: Breast Implant Surgery
- Reconstruction: Reconstruction
  Style 410 Silicone-Filled Breast Implants: Breast Implant Surgery
- Revision-augmentation: Revision-augmentation
  Style 410 Silicone-Filled Breast Implants: Breast Implant Surgery
- Revision-reconstruction: Revision-reconstruction
  Style 410 Silicone-Filled Breast Implants: Breast Implant Surgery
Period: Overall Study
Arm/Group | Augmentation | Reconstruction | Revision-augmentation | Revision-reconstruction
Started | 492 | 225 | 156 | 68
Completed | 375 | 144 | 99 | 43
Not Completed | 117 | 81 | 57 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Augmentation | Reconstruction | Revision-augmentation | Revision-reconstruction | Total
Number analyzed (Participants) | 492 | 225 | 156 | 68 | 941
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 492 | 218 | 156 | 65 | 931
  >=65 years | 0 | 7 | 0 | 3 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 492 | 225 | 156 | 68 | 941
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Local Complications
Description: By patient risk of complications occurring in at least 5% of patients in 1 or more cohorts
Time Frame: 10 years
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Arm/Group | Augmentation | Reconstruction | Revision-augmentation | Revision-reconstruction
Number analyzed (Participants) | 492 | 225 | 156 | 68
Percentage of Patients
  Capsular Contracture | 9.2 [6.7 to 12.6] | 14.5 [10.1 to 20.6] | 11.9 [7.2 to 19.3] | 26.8 [16.8 to 41.1]
  Asymmetry | 1.2 [0.5 to 2.9] | 12.4 [8.4 to 18.1] | 6.9 [3.6 to 13.1] | 17.4 [9.6 to 30.5]
  Breast Pain | 4.5 [2.8 to 7.1] | 8.2 [4.9 to 13.7] | 5.2 [2.3 to 11.5] | 7.8 [2.9 to 20.4]
  Wrinkling/Rippling | 0.9 [0.3 to 2.4] | 6.2 [3.3 to 11.4] | 3.7 [1.5 to 8.6] | 12.8 [6.1 to 25.6]
  Infection | 1.7 [0.8 to 3.3] | 6.1 [3.5 to 10.7] | 2.1 [0.7 to 6.3] | 8.5 [3.6 to 19.5]
  Implant Malposition | 4.7 [3.1 to 7.3] | 5.7 [3.1 to 10.5] | 9.1 [5.2 to 15.6] | 8.0 [3.0 to 20.5]
  Swelling | 4.0 [2.5 to 6.3] | 5.3 [2.8 to 9.7] | 2.7 [1.0 to 7.1] | 3.2 [0.8 to 12.4]
  Seroma/Fluid Accumulation | 1.6 [0.8 to 3.3] | 2.8 [1.1 to 6.6] | 3.2 [1.2 to 8.4] | 6.2 [2.4 to 15.8]

2. Secondary Outcome: Satisfaction With Breast Implants as Determined by Patients and Physicians on a 5-point Scale.
Description: Satisfaction score on a 5-point scale, where 1 is definitely dissatisfied and 5 is definitely satisfied
Time Frame: 10 years
Population: All patients who had a breast implant satisfaction rating
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Augmentation | Reconstruction | Revision-augmentation | Revision-reconstruction
Number analyzed (Participants) | 292 | 134 | 72 | 40
units on a scale
  Physician Satisfaction | 4.8 (0.7) | 4.6 (0.8) | 4.5 (1.0) | 4.4 (0.9)
  Patient Satisfaction | 4.8 (0.7) | 4.6 (0.8) | 4.4 (1.1) | 4.5 (0.9)

ADVERSE EVENTS:
Arm/Group | Augmentation | Reconstruction | Revision-augmentation | Revision-reconstruction
Serious Adverse Events (participants affected / at risk) | 0/492 | 0/225 | 0/156 | 0/68
Other Adverse Events (participants affected / at risk) | 0/492 | 0/225 | 0/156 | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.